CLINICAL TRIAL: NCT00458302
Title: A Randomised, Controlled, Open-label Trial to Compare the Efficacy, Safety and Tolerability of a Treatment Simplification by Darunavir/Ritonavir (DRV/r) 800/100 mg O.D. vs a Triple Combination Therapy With DRV/r in HIV-1 Infected Patients With Undetectable Plasma HIV-RNA on Their Current Treatments.
Brief Title: Treatment Simplification by Darunavir/Ritonavir 800/100 mg Once a Day Versus a Triple Combination Therapy With Darunavir/Ritonavir
Acronym: MONET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR013159; TMC114HIV3006 (Other: Janssen-Cilag International NV); 2006-006437-40 (EudraCT Number)
Record Dates: First submitted 2007-04-06; First posted 2007-04-10 (Estimated); Results first posted 2010-02-26 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: HIV Infections; AIDS Virus; Human Immunodeficiency Virus; Acquired Immunodeficiency Syndrome Virus
Keywords: HIV; Monotherapy; Darunavir; Protease inhibitor; Early pre-treated; Undetectable; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Darunavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- darunavir monotherapy (Experimental): darunavir (DRV, TMC114) 800 mg qd (2 x 400 mg tablet) monotherapy for 144 weeks
  Interventions: Drug: darunavir (DRV, TMC114)
- darunavir + 2 NRTI (Experimental): darunavir (DRV, TMC114) 800 mg qd (2 x 400 mg tablet) + 2 NRTI for 144 weeks
  Interventions: Drug: darunavir (DRV, TMC114)

INTERVENTIONS:
Drug: darunavir (DRV, TMC114) — 800 mg qd (2 x 400 mg tablet) + 2 NRTI for 144 weeks
  Arms: darunavir + 2 NRTI
Drug: darunavir (DRV, TMC114) — 800 mg qd (2 x 400 mg tablet) monotherapy for 144 weeks
  Arms: darunavir monotherapy

SUMMARY:
The purpose of the study is to compare the efficacy, safety and tolerability of darunavir/ritonavir 800/100 mg once a day (O.D.) as a monotherapy versus a triple combination therapy containing 2 nucleosides and darunavir/ritonavir in 250 HIV-1 infected patients who have been on Highly Active Antiretroviral Therapy (HAART) and have plasma viral load below 50 copies/ml for at least 24 weeks.

DETAILED DESCRIPTION:
This study is randomised (patients are assigned different treatments based on chance), controlled, open-label trial to compare the efficacy, safety and tolerability of darunavir/ritonavir (DRV/r) 800/100 mg once a day (O.D.) as a monotherapy versus a triple combination therapy containing 2 nucleosides and DRV/r in 250 HIV-1 infected patients. Patients will be considered eligible if they have not changed any antiretroviral drugs for at least 8 weeks prior to screening and have documented evidence of plasma viral load (or plasma HIV-1 RNA) < 50 copies/mL for at least 24 weeks prior to being screened. The trial will consist of a screening period up to 4 weeks, a 48-week treatment period, followed by a 4-week follow-up (FU) period. The primary objective is to demonstrate non-inferiority in efficacy of DRV/r versus the triple combination therapy containing DRV/r, with respect to confirmed virologic response, defined as plasma HIV-1 RNA < 50 copies/mL at 48 weeks.Patients will be assigned a study medication based on a 1:1 ratio to either switch to a triple combination therapy containing 2 nucleosides and DRV/r 800/100 mg O.D, or initiate monotherapy with DRV/r 800/100 mg O.D. Patients in the triple combination arm who are already on 2 nucleosides prior to randomisation may remain on these or switch them at baseline. Patients randomised to the monotherapy arm will discontinue Highly Active Antiretroviral Therapy (HAART) at baseline and commence DRV/r 800/100 mg O.D. A Data and Safety Monitoring Board (DSMB) has been commissioned for this study. The role of the DSMB is to review the progress of the trial and the accumulating data to detect evidence of early safety issues for the patients while the trial is ongoing. An interim analysis will be performed after 24 weeks of treatment. The results of the Week 24 analysis will be used to determine whether long-term follow-up to 72 and 96 weeks will be done. The protease inhibitor (PI) component of the regimen cannot be changed until the end of the treatment period and the nucleoside reverse transcriptase inhibitors (NRTIs) cannot be modified until the end of the treatment period with the following exception: single antiretroviral (ARV) substitutions will be allowed for tolerability/toxicity reasons, as long as this can be linked to an adverse event (AE) or an serious adverse event (SAE). After withdrawal of the patient from the trial, changes in the ARV regimen are allowed after the assessments of the withdrawal visit have been performed.

Temporary interruption of all ARVs will be allowed in the event of suspected toxicity, as long as the temporary interruption is associated with and can be linked to an AE or a SAE. For the control arm, the nucleoside analogues could be re-optimized at baseline or on study, and all approved ARVs allowed. However, PIs other than DRV/r are not allowed during the treatment period. Patients who cannot resume study medication will have to be withdrawn. A physical examination will be done at protocol-scheduled visits and vital signs will be monitored at each study visit. In addition, at each study visit, every patient will be asked about the occurrence of or change to AEs since they were last seen by the investigator. Laboratory samples for haematology and serum chemistry will be drawn and the results determined and transmitted to the investigator. Urinalysis will be performed. Pregnancy test will be done at each visit for female participants of child-bearing potential. The primary endpoint will be the proportion with virologic response, defined as a confirmed plasma HIV-1 RNA < 50 copies/mL at Week 48.The study hypothesis is that DRV/r monotherapy will be as effective as a triple combination regimen and will be well tolerated in this early pre-treated HIV-1 patients. Two 400mg tablets of darunavir once daily orally within 30 minutes after completion of a meal for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented HIV-1 infection
* Patients currently receiving HAART for at least 24 weeks
* Plasma viral load < 50 copies/mL for at least 24 weeks prior to screening (two results must be documented)
* Patients taking the same antiretroviral combination for at least 8 weeks before screening
* Patients and physician's preference to change the current HAART regimen for reasons of simplification and/or toxicity
* CD4 > 100/mm3 at the start of HAART and > 200/mm3 at screening.

Exclusion Criteria:

* No history of virological failure defined as two consecutive plasma HIV-1 RNA > 500 copies/mL while on previous or current antiretroviral therapy
* No history of any primary PI mutations as defined by the IAS-USA guidelines 2006
* No patients co-infected with hepatitis B
* No pregnant or breastfeeding women
* No active clinically significant disease or life threatening disease or findings during screening of medical history or physical examination that, in the investigator's opinion, would compromise the patient's safety or outcome of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2007-06; Primary Completion 2009-02 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (27):
- Vienna, Austria
- Belgium (2):
  - Antwerp
  - Brussels
- Denmark (4):
  - Aarhus
  - Copenhagen
  - Hvidovre
  - Odense
- Germany (5):
  - Berlin
  - Frankfurt
  - Hamburg
  - Hanover
  - Kÿln N/A
- Budapest, Hungary
- Israel (3):
  - Jerusalem
  - Tel Aviv
  - Tel Litwinsky
- Portugal (2):
  - Lisbon
  - Porto
- Russia (2):
  - Moscow
  - Saint Petersburg
- Spain (5):
  - Barcelona
  - Donostia Guipuzcoa
  - Granada
  - Madrid
  - Valladolid
- Sankt Gallen, Switzerland
- London, United Kingdom

REFERENCES:
- [Derived] Arribas JR, Horban A, Gerstoft J, Fatkenheuer G, Nelson M, Clumeck N, Pulido F, Hill A, van Delft Y, Stark T, Moecklinghoff C. The MONET trial: darunavir/ritonavir with or without nucleoside analogues, for patients with HIV RNA below 50 copies/ml. AIDS. 2010 Jan 16;24(2):223-30. doi: 10.1097/QAD.0b013e3283348944. PMID 20010070

RESULTS

PARTICIPANT FLOW:
Recruitment Details: xxxxx
Groups:
- DRV/r+2NRTIs: 800 mg qd (2 x 400 mg tablet) + 2 NRTI for 144 weeks
- DRV/r: 800 mg qd (2 x 400 mg tablet) monotherapy for 144 weeks
Period: Overall Study
Arm/Group | DRV/r+2NRTIs | DRV/r
Started | 129 | 127
Completed | 109 | 103
Not Completed | 20 | 24
Not completed — Adverse Event | 4 | 14
Not completed — Pregnancy | 2 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Inc/Exc Criteria Not Met | 1 | 1
Not completed — Study Termination By Sponsor | 1 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Other | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DRV/r+2NRTIs | DRV/r | Total
Number analyzed (Participants) | 129 | 127 | 256
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 128 | 125 | 253
  >=65 years | 1 | 2 | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 44.1 (9.74) | 43.4 (9.14) | 43.7 (9.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 28 | 50
  Male | 107 | 99 | 206
Region of Enrollment [Number; unit: participants]
  AUSTRIA | 9 | 7 | 16
  BELGIUM | 12 | 12 | 24
  DENMARK | 14 | 14 | 28
  GERMANY | 14 | 14 | 28
  HUNGARY | 6 | 5 | 11
  ISRAEL | 1 | 7 | 8
  ITALY | 11 | 5 | 16
  POLAND | 9 | 20 | 29
  PORTUGAL | 7 | 7 | 14
  RUSSIAN FEDERATION | 9 | 2 | 11
  SPAIN | 24 | 24 | 48
  SWITZERLAND | 1 | 1 | 2
  UNITED KINGDOM | 12 | 9 | 21
plasma viral load [Number; unit: participants] — plasma viral load (HIV-1 RNA copies/ml)
  participants
    < 50 | 125 | 118 | 243
    50-400 | 4 | 7 | 11
    400-1000 | 0 | 0 | 0
    > 1000 | 0 | 2 | 2
CD4+ cell count (absolute count) [Median (Full Range); unit: cells/µl] | 579.0 [163 to 1888] | 571.0 [162 to 1451] | 573.5 [162 to 1888]

OUTCOME MEASURES:

1. Primary Outcome: Virological Response [Per Protocol (PP) - Time to Loss of Virologic Response (TLOVR), < 50 Copies/ml, Week 48]
Description: Virological response is defined as the number of patients in the PP population with a plasma viral load < 50 HIV RNA copies/ml at Week 48. Treatment failure was defined as two consecutive HIV RNA levels ≥ 50 copies/mL, or discontinuation of randomised treatment (known as TLOVR). In addition, any switch in background nucleoside reverse transcriptase inhibitors (NRTIs) equaled failure* (referred to as a Switch Equals Failure analysis). *Discontinuations and rechallenge with NRTIs are taken into account until Week 48
Time Frame: Week 48
Population: PP population: all randomised patients who took study drug, and who did not deviate from the protocol.This excludes 10 patients with major protocol deviations.
Measure: Number; unit: participants
Arm/Group | DRV/r+2NRTIs | DRV/r
Number analyzed (Participants) | 123 | 123
participants | 108 | 106
Statistical Analysis 1: Comparison: DRV/r+2NRTIs vs DRV/r; Assuming a virologic response rate of 90% at 48 weeks for both treatment arms, 111 patients were required per treatment arm to establish non-inferiority of DRV/r versus triple regimen with a maximum allowable difference of 12%, with a one-sided significance level of p=0.025 and 80% power. To account for a maximum of 10% major protocol violations that would be excluded from the on-protocol analysis, 125 patients were recruited in each treatment arm, so 250 patients in total; Test type: Non-Inferiority or Equivalence — The primary comparison was performed at Week 48. If at Week 48, the lower limit of the 95% two-sided confidence interval of the difference between DRV/r and DRV/r+2NRTIs exceeds -12%, non-inferiority of the DRV/r 800/100 once a day (O.D) monotherapy versus the DRV/r 800/100 mg O.D. plus two NRTIs triple combination therapy was concluded; Difference in proportion of response = -1.6, 95% CI 2-sided [-10.1 to 6.8] — Difference in proportion of response DRV/r minus DRV/r+2NRTIs

2. Secondary Outcome: Virological Response [Intent To Treat (ITT) - TLOVR, < 50 Copies/ml, Week 48]
Description: Virological response is defined as the number of patients in the ITT population with a plasma viral load < 50 HIV RNA copies/ml at Week 48. Treatment failure was defined as two consecutive HIV RNA levels ≥ 50 copies/mL, or discontinuation of randomised treatment (known as TLOVR). In addition, any switch in background nucleoside reverse transcriptase inhibitors (NRTIs) equaled failure* (referred to as a Switch Equals Failure analysis). *Discontinuations and rechallenge with NRTIs are taken into account until start of Week 48 window
Time Frame: Week 48
Population: ITT population: all randomised patients who took study drug, regardless of their compliance with the protocol.
Measure: Number; unit: participants
Arm/Group | DRV/r+2NRTIs | DRV/r
Number analyzed (Participants) | 129 | 127
participants | 110 | 107
Statistical Analysis 1: Comparison: DRV/r+2NRTIs vs DRV/r; Assuming a virologic response rate of 90% at 48 weeks for both treatment arms, 111 patients were required per treatment arm to establish non-inferiority of DRV/r versus triple regimen with a maximum allowable difference of 12%, with a one-sided significance level of p=0.025 and 80% power. To account for a maximum of 10% major protocol violations that would be excluded from the on-protocol analysis, 125 patients were recruited in each treatment are, so 250 patients in total; Test type: Non-Inferiority or Equivalence — If at Week 48, the lower limit of the 95% two-sided confidence interval of the difference between DRV/r and DRV/r+2NRTIs exceeds -12%, non-inferiority of the DRV/r 800/100 once a day (O.D) monotherapy versus the DRV/r 800/100 mg O.D. plus two NRTIs triple combination therapy was concluded; Difference in proportion of response = -1.0, 95% CI 2-sided [-9.9 to 7.8] — Difference in proportion of response DRV/r minus DRV/r+2NRTIs

3. Secondary Outcome: Virological Response [Per Protocol (PP), TLOVR - Switch Equals Failure, < 50 Copies/ml, Week 144]
Description: Virological response is defined as the number of patients in the PP population with a plasma viral load < 50 HIV RNA copies/ml at Week 144. Treatment failure was defined as two consecutive HIV RNA levels ≥ 50 copies/mL, or discontinuation of randomised treatment (known as TLOVR). In addition, any switch in background nucleoside reverse transcriptase inhibitors (NRTIs) equaled failure* (referred to as a Switch Equals Failure analysis). *Discontinuations and rechallenge with NRTIs are taken into account until Week 144
Time Frame: Week 144
Population: PP population: all randomised subjects who took study drug, and who did not deviate from the protocol.This excludes 13 subjects with major protocol deviations.
Measure: Number; unit: participants
Arm/Group | DRV/r+2NRTIs | DRV/r
Number analyzed (Participants) | 121 | 122
participants | 94 | 88

4. Secondary Outcome: Virological Response [Intent To Treat (ITT), TLOVR - All Switches Included, < 50 Copies/ml, Week 144]
Description: Virological response is defined as the number of patients in the ITT population with a plasma viral load < 50 HIV RNA copies/ml at Week 144. Treatment failure was defined as two consecutive HIV RNA levels ≥ 50 copies/mL, or discontinuation of randomised treatment (known as TLOVR). All switches included means that all data even after any changes of treatment were kept. *Discontinuations and rechallenge with NRTIs are taken into account until start of Week 144 window.
Time Frame: Week 144
Population: ITT population: all randomised patients who took study drug, regardless of their compliance with the protocol.
Measure: Number; unit: participants
Arm/Group | DRV/r+2NRTIs | DRV/r
Number analyzed (Participants) | 129 | 127
participants | 106 | 106
Statistical Analysis 1: Comparison: DRV/r+2NRTIs vs DRV/r; Test type: Superiority or Other; Difference in proportion of response = 1.29, 95% CI 2-sided [-7.99 to 10.58] — Difference in proportion of response DRV/r minus DRV/r+2NRTIs

5. Secondary Outcome: Virological Response [Per Protocol (PP), TLOVR - Switch Equals Failure, <200 Copies/ml, Week 144]
Description: Virological response is defined as the number of patients in the PP population with a plasma viral load < 200 HIV RNA copies/ml at Week 144. Treatment failure was defined as two consecutive HIV RNA levels ≥ 50 copies/mL, or discontinuation of randomised treatment (known as TLOVR). In addition, any switch in background nucleoside reverse transcriptase inhibitors (NRTIs) equaled failure* (referred to as a Switch Equals Failure analysis). *Discontinuations and rechallenge with NRTIs are taken into account until Week 144
Time Frame: week 144
Population: PP population: all randomised patients who took study drug, and who did not deviate from the protocol. This excludes 13 patients with major protocol deviations.
Measure: Number; unit: Participants
Arm/Group | DRV/r+2NRTIs | DRV/r
Number analyzed (Participants) | 121 | 122
Participants | 102 | 95

6. Secondary Outcome: Mean Change From Baseline in CD4+ Cell Count
Description: The mean change in CD4+ cell count from baseline was calculated with a last observation carried forward method; i.e. the last observed value was carried forward, irrespective of the reason for discontinuation.
Time Frame: at week 4, 12, 24, 36, 48, 60, 72, 84, 96, 112, 128, 144
Population: ITT: all randomized patients who had at least 1 dose of study medication, regardless of their adherence to the protocol
Measure: Mean (Standard Error); unit: number of cells/L (x10^6)
Arm/Group | DRV/r+2NRTIs | DRV/r
Number analyzed (Participants) | 129 | 127
number of cells/L (x10^6)
  week 4 | -16.9 (15.7) | -32.9 (14.6)
  week 12 | -23.6 (14.7) | -20.7 (15.2)
  week 24 | -5.4 (14.6) | -35.8 (14.2)
  week 36 | -1.2 (15.8) | -21.1 (14.3)
  week 48 | -19.0 (14.7) | -15.1 (16.0)
  week 60 | -4.0 (14.9) | -2.3 (14.4)
  week 72 | 24.1 (16.1) | -12.3 (14.3)
  week 84 | 34.6 (17.2) | -3.7 (15.0)
  week 96 | 49.1 (15.9) | 54.8 (16.2)
  week 112 | 106.0 (16.7) | 87.5 (16.2)
  week 128 | 117.3 (18.3) | 90.4 (14.9)
  week 144 | 99.3 (15.7) | 94.9 (15.0)

7. Secondary Outcome: Resistance Determinations
Description: Number of patients with resistance mutations at any time point when a patient had a viral load > 50 copies/mL after randomization.
Time Frame: at each visit from baseline to week 144
Population: ITT: all randomised patients who had at least 1 dose of study medication, regardless of their adherence to the protocol.
Measure: Number; unit: number of participants
Arm/Group | DRV/r+2NRTIs | DRV/r
Number analyzed (Participants) | 129 | 127
number of participants
  >= 1 HIV-1 RNA > 50 copies/mL | 42 | 48
  >= 1 successful genotype after baseline | 23 | 31
  >= 1 IAS-USA primary PI mutations | 1 | 1
  >= 1 DRV RAMs | 0 | 1
  NRTI RAMs | 1 | 0
  M184V mutation | 1 | 0
  no primary PI, DRV, NRTI or M184 V mutations | 22 | 30

8. Secondary Outcome: Change From Baseline in Health-Related Quality of Life - FAHI Questionnaire Total Score
Description: The FAHI is a validated health-related quality of life questionnaire. The questionnaire consist of 44 items and includes 5 functional scales (physical, social, emotional, functional and global well-being and cognitive function). Each item is assessing the impact of HIV on a scale from 0 (not at all) to 5 (very much).
Time Frame: at baseline, week 48, 96 and 144
Population: ITT: all randomised patients who had at least 1 dose of study medication, regardless of protocol adherence. A LOCF method was used for calculation.
Measure: Mean (Standard Error); unit: points on a scale
Arm/Group | DRV/r+2NRTIs | DRV/r
Number analyzed (Participants) | 126 | 112
points on a scale
  week 48 | 1.7 (1.7) | 1.7 (2.0)
  week 96 | 0.4 (1.6) | 3.5 (2.4)
  week 144 | 0.7 (1.7) | 3.1 (2.4)

9. Secondary Outcome: Change From Baseline in Health-Related Quality of Life - FAHI Questionnaire Cognitive Function Subscale
Description: The FAHI cognitive function subscale. Each item is assessing the impact of HIV on cognitive function on a scale from 0 (not at all) to 5 (very much).
Time Frame: at baseline, week 48, 96 and 144
Population: as for outcome 8
Measure: Mean (Standard Error); unit: points on a scale
Arm/Group | DRV/r+2NRTIs | DRV/r
Number analyzed (Participants) | 127 | 115
points on a scale
  week 48 | 0.1 (0.2) | -0.1 (0.2)
  week 96 | -0.1 (0.2) | -0.1 (0.2)
  week 144 | 0.1 (0.2) | -0.1 (0.2)

10. Secondary Outcome: Change From Baseline in Health-Related Quality of Life - FAHI Questionnaire Emotional Well-Being Subscale
Description: The FAHI emotional well-being subscale. Each item is assessing the impact of HIV on emotional well-being on a scale from 0 (not at all) to 5 (very much).
Time Frame: at baseline, week 48, 96 and 144
Population: as for outcome 8
Measure: Mean (Standard Error); unit: points on a scale
Arm/Group | DRV/r+2NRTIs | DRV/r
Number analyzed (Participants) | 128 | 118
points on a scale
  week 48 | 0.1 (0.6) | 1.8 (0.7)
  week 96 | 1.0 (0.5) | 1.3 (0.7)
  week 144 | 1.4 (0.5) | 1.7 (0.7)

11. Secondary Outcome: Change From Baseline in Health-Related Quality of Life - FAHI Questionnaire Functional and Global Well-Being Subscale
Description: The FAHI functional and global well-being subscale. Each item is assessing the impact of HIV on functional and global well-being on a scale from 0 (not at all) to 5 (very much).
Time Frame: at baseline, week 48, 96 and 144
Population: as for outcome 8
Measure: Mean (Standard Error); unit: points on a scale
Arm/Group | DRV/r+2NRTIs | DRV/r
Number analyzed (Participants) | 127 | 116
points on a scale
  week 48 | 0.3 (0.8) | -0.8 (0.7)
  week 96 | -0.1 (0.7) | 0.4 (0.9)
  week 144 | -0.6 (0.8) | 0.0 (1.0)

12. Secondary Outcome: Change From Baseline in Health-Related Quality of Life - FAHI Questionnaire Physical Well-Being Subscale
Description: The FAHI physical well-being subscale. Each item is assessing the impact of HIV on physical well-being on a scale from 0 (not at all) to 5 (very much).
Time Frame: at baseline, week 48, 96 and 144
Population: as for outcome 8
Measure: Mean (Standard Error); unit: points on a scale
Arm/Group | DRV/r+2NRTIs | DRV/r
Number analyzed (Participants) | 128 | 118
points on a scale
  week 48 | 0.6 (0.5) | 1.0 (0.8)
  week 96 | 0.4 (0.5) | 1.4 (0.9)
  week 144 | 0.0 (0.5) | 1.0 (0.8)

13. Secondary Outcome: Change From Baseline in Health-Related Quality of Life - FAHI Questionnaire Social Well-Being Subscale
Description: The FAHI social well-being subscale. Each item is assessing the impact of HIV on physical well-being on a scale from 0 (not at all) to 5 (very much).
Time Frame: at baseline, week 48, 96 and 144
Population: as for outcome 8
Measure: Mean (Standard Error); unit: points on a scale
Arm/Group | DRV/r+2NRTIs | DRV/r
Number analyzed (Participants) | 126 | 115
points on a scale
  week 48 | 0.4 (0.5) | -0.2 (0.5)
  week 96 | -0.6 (0.5) | 0.8 (0.6)
  week 144 | -0.3 (0.5) | 0.6 (0.6)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study. Mean exposure at the time of primary analysis (Week 48) was 457.3 days for the overall study population (462.3 days for the DRV/r+2NRTIs group and 452.2 days for the DRV/r group).
Description: Adverse events were either reported by the subjects voluntarily or were obtained by means of interviewing subjects in a non-directed manner at study visits.
Arm/Group | DRV/r+2NRTIs | DRV/r | Total
Serious Adverse Events (participants affected / at risk) | 14/129 | 14/127 | 28/256
Other Adverse Events (participants affected / at risk) | 98/129 | 103/127 | 201/256
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DRV/r+2NRTIs (N=129) | DRV/r (N=127) | Total (N=256)
Gastroenteritis (Infections and infestations) | 1 | 0 | 1
Hepatitis A (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 1
Subcutaneous Abscess (Infections and infestations) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1
Hepatitis C (Infections and infestations) | 0 | 1 | 1
Neurosyphilis (Infections and infestations) | 0 | 2 | 2
Secondary Syphilis (Infections and infestations) | 0 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Hodgkin's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Tongue Neoplasm Malignant Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0 | 1
Nervous System Disorder (Nervous system disorders) | 1 | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0 | 1
Duodenal Ulcer (Gastrointestinal disorders) | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 1 | 1 | 2
Aspartate Aminotransferase Increased (Investigations) | 1 | 0 | 1
Csf Pressure Decreased (Investigations) | 0 | 1 | 1
Lipase Increased (Investigations) | 0 | 1 | 1
Somatoform Disorder (Psychiatric disorders) | 1 | 0 | 1
Psychotic Disorder (Psychiatric disorders) | 0 | 2 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1
Cataract Operation (Surgical and medical procedures) | 1 | 0 | 1
Varicose Vein Operation (Surgical and medical procedures) | 0 | 1 | 1
Uveitis (Eye disorders) | 0 | 1 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1 | 1
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Incisional Hernia (Injury, poisoning and procedural complications) | 0 | 1 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 1 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DRV/r+2NRTIs (N=129) | DRV/r (N=127) | Total (N=256)
Diarrhoea (Gastrointestinal disorders) | 26 | 26 | 52
Vomiting (Gastrointestinal disorders) | 9 | 1 | 10
Nausea (Gastrointestinal disorders) | 7 | 5 | 12
Bronchitis (Infections and infestations) | 12 | 10 | 22
Nasopharyngitis (Infections and infestations) | 10 | 15 | 25
Respiratory Tract Infection (Infections and infestations) | 9 | 1 | 10
Upper Respiratory Tract Infection (Infections and infestations) | 7 | 12 | 19
Haematuria (Renal and urinary disorders) | 12 | 7 | 19
Leukocyturia (Renal and urinary disorders) | 7 | 6 | 13
Headache (Nervous system disorders) | 10 | 12 | 22
Hypertension (Vascular disorders) | 9 | 6 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 7 | 15
Depression (Psychiatric disorders) | 7 | 12 | 19
Fatigue (General disorders) | 6 | 7 | 13
Hypercholesterolaemia (Metabolism and nutrition disorders) | 6 | 19 | 25
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 8 | 12
Rash (Skin and subcutaneous tissue disorders) | 4 | 8 | 12
Blood Cholesterol Increased (Investigations) | 2 | 7 | 9

LIMITATIONS AND CAVEATS:
This study was not blinded and not designed to demonstrate a safety benefit to stopping nucleoside analogues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor (SP) shall have the 1st right to present the Data without approval from the Principal Investigator (PI). If no publication is submitted by SP within 12 months after closure, or after SP confirms there will be no publication, the PI shall have the right to publish. Prior to submission, the PI will provide the SP with at least 45 days for review of a manuscript. If requested, the PI will withhold such publication for up to an additional 60 days to allow for filing of a patent application